CLINICAL TRIAL: NCT06318013
Title: Comparison of Perineural and Systemic Dexamethasone Use in Third Molar Dental Surgeries in Terms of Anesthesia Duration and Postoperative Complaints: a Controlled, Randomized Observational Study.
Brief Title: Perineural and Systemic Dexamethasone Use in Dental Surgeries in Terms of Anesthesia Duration and Postop Complaints
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Dogan Ilgaz Kaya, Assistant Professor, Karamanoğlu Mehmetbey University
Other Study IDs: 2022-KAEK-15427-04-204-2022101
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Impacted Third Molar Tooth
Keywords: Impacted third molar; Dexamethasone; anesthesia duration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Group receiving only local anesthesia
  Interventions: Diagnostic Test: vitality test
- Intravenous Dexamethasone: Group using dexamethasone IV
  Interventions: Diagnostic Test: vitality test
- Perineural Dexamethasone: group administered perineural dexamethasone
  Interventions: Diagnostic Test: vitality test

INTERVENTIONS:
Diagnostic Test: vitality test — A vitality test will be performed using a vitalometer to check if the drowsiness is gone

SUMMARY:
Participants will be asked to use some medications after the tooth extraction procedure. These drugs can be used in different ways. Investigators plan to monitor the pain, swelling and duration of anesthesia in the body as a result of participants use.

DETAILED DESCRIPTION:
PURPOSE OF THE RESEARCH: Third molar tooth extraction is a frequently performed procedure in dentistry. Depending on the degree of impaction of the teeth, this procedure causes postoperative sequelae such as pain and edema that reduce the quality of life. Clinical studies have proven that the use of antibiotics, physiotherapy, corticosteroid treatment, and antiseptic mouthwashes reduce postoperative complications.

There are different ways to use costosteroids in dental practice. Intravenous, intramuscular, perineural and oral tablet administration are the most preferred. It has been proven that if dexamethasone is given systemically, the duration of anesthesia in shoulder surgeries is prolonged and post-operative pain is less. (1) However, no study evaluating this parameter regarding twenty-year-old surgeries has been found in the literature. The aim of this study is to compare the post-procedure numbness duration and postoperative sequelae in patients who were administered dexamethasone intravenously and perineurally perioperatively.

Material Method: The study is planned to be carried out at Karamanoğlu Mehmetbey University Ahmet Keleşoğlu Faculty of Dentistry. Patients who apply to the Oral and Maxillofacial Surgery Department for impacted wisdom tooth extraction and are directed to the local intervention room for tooth extraction will be asked whether they want to participate in the study after leaving the procedure room. Patients who want to participate in the study will have an informed consent form read and their signature will be taken if they declare that they want to participate in the study. Patients participating in the study will be checked for drowsiness every 30 minutes for the first 2 hours after the procedure, and every 15 minutes from the 3rd hour onwards. Drowsiness control will be done with a device called vitalometer that measures the vitality of teeth. The start time of the operation and the time the numbness subsides will be recorded. On the 1st, 3rd and 7th days following the operation, tragus-pogonion, tragus-mouth canthus and gonion-lateral canthus will be measured to evaluate swelling. Measurement will be made with a tape measure. Additionally, pain assessment and maximum mouth opening measurement will be performed with a visual analog scale on the same days. Manual caliper will be used for mouth opening measurement.

The inclusion criteria for the study were patients between the ages of 18 and 35, with ASA class 1, impacted teeth in Class II position B according to the Pell and Gregory classification, and without signs of inflammation and dental pathology. Pregnant or breastfeeding women, patients with diabetes, endocrine diseases, hypertension patients, bleeding disorders or patients using anticoagulants will be excluded from the study. If the duration of the surgical procedure is more than 30 minutes, if repeated doses of local anesthetic are injected during the procedure, and if surgical complications occur during the procedure, patients will be excluded from the study. This information will be checked from the epicrisis report filled out by the physician performing the operation.

Three groups will be formed by examining the procedures applied to the patients and the medications given to them from the patient follow-up program of the faculty of dentistry. It is planned to include 20 patients in each group. These are those who were administered perineural dexamethasone, those who were administered intravenous dexamethasone, and those who were not administered dexamethasone (control). The results obtained from the measurements will be compared in these 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1, impacted teeth in Class II position B according to the Pell and Gregory classification, with no signs of inflammation and no dental pathology

Exclusion Criteria:

* Pregnant or breastfeeding women, patients with diabetes, endocrine disease, hypertension patients, patients with bleeding disorders or using anticoagulants

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, male and female patients between the ages of 18-35
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
Swelling | 1 week
  In order to determine the course of postoperative edema in patients with tooth extraction, tragus-pogonion (S1), tragus-mouth canthus (S2) and gonion-lateral canthus (S3) will be measured with the help of a tape measure.
Duration of anesthesia | 6 hours
  After anesthesia, the time it takes for numbness to subside will be measured in minutes. A vitalometer device will be used to check that anesthesia has passed.

SECONDARY OUTCOMES:
Pain Score | 1 week
  Vas scale (no pain:0-intolerable pain:10) will be used to measure postoperative pain in patients with tooth extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Aktı, Dr, Principal Investigator — Selcuk University
Locations (1):
- Karamanoğlu Mehmetbey University Ahmet Keleşoğlu Faculty of Dentistry, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not need to record participants' personal data for this study.

REFERENCES:
- [Result] Ruthvik S, Krishnan M, George M, Kumar SP, Lakshmanan S. Efficacy of Dexamethasone Diluted Saline Irrigant on Postoperative Sequelae in Patients Undergoing Lower Third Molar Surgery: A Prospective Clinical Study. Cureus. 2023 Sep 18;15(9):e45436. doi: 10.7759/cureus.45436. eCollection 2023 Sep. PMID 37859912
- [Result] Poorna P, Shetty P, Kalyani V, Shetty S, Upadya M, Mithra P. A comparative evaluation of the effect of addition of 8 mg dexamethasone to 2% lignocaine with adrenaline in mandibular third molar surgery: a split mouth randomised double blind study. Front Oral Health. 2024 Feb 9;5:1349832. doi: 10.3389/froh.2024.1349832. eCollection 2024. PMID 38404531
- [Result] Priyanga R, Balamurugan R, Rajan PS. Comparison of dexamethasone administration through sublingual and intramuscular routes for evaluation of pain, swelling, and trismus after impacted mandibular third molar surgery-a prospective randomized controlled study. Oral Maxillofac Surg. 2022 Mar;26(1):155-159. doi: 10.1007/s10006-021-00978-4. Epub 2021 Jun 5. PMID 34091813
- [Derived] Kaya DI, Akti A. Comparison of perineural and systemic dexamethasone use in impacted third molar surgeries in terms of anesthesia duration and postoperative complaints: a controlled, randomized observational study. BMC Oral Health. 2024 Jun 18;24(1):706. doi: 10.1186/s12903-024-04483-4. PMID 38890655